CLINICAL TRIAL: NCT01800890
Title: Investigating the Safety and Performance of New 2-piece Ostomy Product Concept Compared With SenSura Click in Subjects With Ileostomy
Brief Title: Safety and Performance of New 2-piece Ostomy Product Concept Compared With SenSura Click in Subjects With Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP234
Record Dates: First submitted 2013-02-22; First posted 2013-02-28 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Subjects With an Ileostomy
Keywords: stoma ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment sequence 1 (Other): Subjects randomised to Treatment sequence 1 will test three different products:
  1. Coloplast A
  2. Coloplast B
  3. SenSura Click
  The subjects test the three test products in a randomized order: ABS; BSA, SAB
  Interventions: Device: Coloplast A; Device: Coloplast B; Device: SenSura Click
- Treatment sequence 2 (Experimental): Subjects randomised to Treatment sequence 2 will test three different products:
  1. Coloplast C (C)
  2. Coloplast B (B)
  3. SenSura Click (S)
  The subjects test the three test products in a randomized order: CBS; BSC, SCB
  Interventions: Device: Coloplast B; Device: Coloplast C; Device: SenSura Click
- Treatment sequence 3 (Experimental): Subjects randomised to Treatment sequence 3 will test three different products:
  1. Coloplast A (A)
  2. Coloplast C (C)
  3. SenSura Click (S)
  The subjects test the three test products in a randomized order: ACS; CSA, SAC
  Interventions: Device: Coloplast A; Device: Coloplast C; Device: SenSura Click

INTERVENTIONS:
Device: Coloplast A — Coloplast A is a newly developed 2-piece ostomy appliance
  Arms: Treatment sequence 1; Treatment sequence 3
Device: Coloplast B — Coloplast B is a newly developed 2-piece ostomy appliance
  Arms: Treatment sequence 1; Treatment sequence 2
Device: Coloplast C — Coloplast C is a newly developed 2-piece ostomy appliance
  Arms: Treatment sequence 2; Treatment sequence 3
Device: SenSura Click — The comparator product is the commercial and CE-marked SenSura Click (2-piece) manufactured by Coloplast A/S.

SUMMARY:
The aim of the current clinical investigation is to evaluate the performance and safety of new 2-piece ostomy product concepts.

DETAILED DESCRIPTION:
The new products have been developed to reduce the degree of leakage and other problems related to ostomy appliances in people with a stoma.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority form.
2. Be at least 18 years of age and have full legal capacity.
3. Be able to handle the appliances themselves
4. Have an ileostomy with a diameter between 15 and 40 mm.
5. Have had their ostomy for at least three months.
6. Use minimum 1 baseplate every third day.
7. Currently use 2-piece flat mechanical coupling product with open bag and a coupling size in the inter val of 43-55mm (both extremes included)
8. Must be able to use custom cut product
9. Accept to test three 2-piece products within the study.
10. Negative result of a pregnancy test for women of childbearing age.

Exclusion Criteria:

1. Use irrigation during the study (flush the stoma with water).
2. Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
3. Currently receiving or have within the past month received local or systemic steroid treatment in the peristomal area.
4. Are pregnant or breastfeeding.
5. Participating in other interventional clinical investigations or have previously participated in this investigation.
6. More than three days wear time as usual change pattern.
7. Currently using ostomy belt
8. Currently using extended wear product (Sensura Xpro, Assura TERA, Dansac NovaLife X3, Hollister Flextend, Convatec Durahesive)
9. Have a loop ileostomy
10. Known hypersensitivity towards any of the test products
11. Suffer from peristomal skin problems that preclude participation in the investigation (assessed by the investigation nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, MSc, Study Chair — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject were recruited through the Coloplast user data base.
Pre-assignment Details: Thirty-one subjects signed the informed consent, but 2 subjects were screen failures and did not test any products. These two subjects are not included in the participant flow below.
Groups:
- Test A/ Test B/ SenSura: The subjects first tested Coloplast test product A then Cololpast test product B and finally the comparator SenSura
- Test A/ Test C/ SenSura: The subjects first tested Coloplast test product A then Cololpast test product C and finally the comparator SenSura
- Test B/ SenSura/ Test A: The subjects first tested Coloplast test product B then the comparator SenSura and finally Cololpast test product A
- Test B/ SenSura/ Test C: The subjects first tested Coloplast test product B then the comparator SenSura and finally Cololpast test product C
- Test C/ Test B/ SenSura: The subjects first tested Coloplast test product C then Cololpast test product B and finally the comparator SenSura
- Test C/ SenSura/ Test A: The subjects first tested Coloplast test product C then the comparator SenSura and finally Cololpast test product A
- SenSura/Test A/Test B: The subjects first tested the comparator product SenSura then Coloplast test product A and finally Cololpast test product B
- SenSura/Test A/Test C: The subjects first tested the comparator product SenSura then Coloplast test product A and finally Cololpast test product C
- SenSura/Test C/Test B: The subjects first tested the comparator product SenSura then Coloplast test product C and finally Cololpast test product B
Period: Test Period 1
Arm/Group | Test A/ Test B/ SenSura | Test A/ Test C/ SenSura | Test B/ SenSura/ Test A | Test B/ SenSura/ Test C | Test C/ Test B/ SenSura | Test C/ SenSura/ Test A | SenSura/Test A/Test B | SenSura/Test A/Test C | SenSura/Test C/Test B
Started | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 4 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Test Period 2
Arm/Group | Test A/ Test B/ SenSura | Test A/ Test C/ SenSura | Test B/ SenSura/ Test A | Test B/ SenSura/ Test C | Test C/ Test B/ SenSura | Test C/ SenSura/ Test A | SenSura/Test A/Test B | SenSura/Test A/Test C | SenSura/Test C/Test B
Started | 3 | 3 | 3 | 2 | 4 | 4 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 4 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 3
Arm/Group | Test A/ Test B/ SenSura | Test A/ Test C/ SenSura | Test B/ SenSura/ Test A | Test B/ SenSura/ Test C | Test C/ Test B/ SenSura | Test C/ SenSura/ Test A | SenSura/Test A/Test B | SenSura/Test A/Test C | SenSura/Test C/Test B
Started | 3 | 3 | 3 | 2 | 4 | 4 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 4 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only includes the ITT population. The two screen failures and the subject who did not complete the Test B period as planned are not included.
  The subject that did not complete the test B period was also a screen failure, however it was first discovered after applying a product. Thus, no endpoint data has been recorded for this subject.
Groups:
- Overall Study Population: baseline data is given for subjects in the ITT population
Arm/Group | Overall Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage is assessed using a 4 point leakage scale developed by Coloplast A/S.
  The 4-point leakage scale has four choices
  1. No leakage
  2. Starting to leakage
  3. Leakage
  4. Sudden leakage
  Leakage was assessed at every baseplate change
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Coloplast Test Product A; Coloplast Test Product B; Coloplast Test Product C: new test product
- SenSura: The comparator
Arm/Group | Coloplast Test Product A | Coloplast Test Product B | Coloplast Test Product C | SenSura
Number analyzed (Participants) | 19 | 18 | 18 | 27
Number analyzed (baseplates) | 91 | 83 | 92 | 117
units on a scale | 1.8 (0.7) | 1.8 (0.7) | 1.9 (0.9) | 1.7 (0.8)

ADVERSE EVENTS:
Description: The safety population included all subjects who had signed the informed consent form and had applied at least one product. Thus, 29 subjects were included in the safety population, which included the subjects who anly tested Test B very shortly.
Groups:
- Coloplast Test Product A: Coloplast Test product A is a new test product
- Coloplast Test Product B: Coloplast Test product B is a new test product
- Coloplast Test Product C: Coloplast Test product C is a new test product
- SenSura: The comparator was the CE-marked product SenSura Click
Arm/Group | Coloplast Test Product A | Coloplast Test Product B | Coloplast Test Product C | SenSura
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 1/28
Other Adverse Events (participants affected / at risk) | 6/19 | 8/19 | 4/19 | 6/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product A (N=19) | Coloplast Test Product B (N=19) | Coloplast Test Product C (N=19) | SenSura (N=28)
stenosis of catherter in the right kidney (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product A (N=19) | Coloplast Test Product B (N=19) | Coloplast Test Product C (N=19) | SenSura (N=28)
peristomal skin irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 4 (4) | 4 (5)
stinging skin by fistel (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cramps in the right kidney with sever pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — not related to the product
influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cold (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
bladder infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
peristomal skin irritaion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diarre due to food intolerance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes